CLINICAL TRIAL: NCT05282446
Title: A Phase 1B Study to Examine the Pharmacokinetic and Pharmacodynamic Effects of INV-202 in Subjects With Metabolic Syndrome as Defined by Hypertriglyceridemia, Abdominal Obesity, and Impaired Glucose Tolerance Over 28 Days
Brief Title: A Study to Explore the PK and PD of INV-202 in Metabolic Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inversago Pharma Inc. (Industry)
Responsible Party: Sponsor
Organization: Novo Nordisk A/S (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INV-202 CL-105
Record Dates: First submitted 2022-02-16; First posted 2022-03-16 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INV-202 (Experimental): INV-202 25mg by mouth once daily
  Interventions: Drug: INV-202
- Placebo (Placebo Comparator): Matching placebo by mouth once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: INV-202 — tablet
  Arms: INV-202
Drug: Placebo — matching tablet
  Arms: Placebo

SUMMARY:
INV-202-CL-105 is a phase 1B study to examine the safety and tolerability, as well as the pharmacokinetics (PK) pharmacodynamic (PD) effects of INV-202 in subjects with metabolic syndrome over 28 days.

DETAILED DESCRIPTION:
INV-202-CL-105 is a phase 1B study to examine the safety and tolerability, as well as the pharmacokinetics (PK) pharmacodynamic (PD) effects of INV-202 in subjects with metabolic syndrome over 28 days.

Subjects with metabolic syndrome as defined as an increased waist circumference, hypertriglyceridemia, and glucose intolerance will be randomized to INV-202 or placebo for 28 to assess PK/PD relationships and other biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of a signed and dated informed consent form (ICF).
2. Willing and able to comply with all study procedures for the duration of the study.
3. Male or female, ≥18 and ≤65 years of age.
4. Waist circumference ≥88 cm for female subjects or ≥102 cm for male subjects.
5. Fasting triglyceride >1.5 mmol/L for males and females.
6. An OGTT indicating impaired glucose tolerance as indicated by a 2-hour value >140 mg/dl or any value >200 mg/dl at any time point or a HbA1C level ≥5.7% but ≤6.4%.

Exclusion Criteria:

1. Female who is lactating at screening.
2. Female who is pregnant according to a pregnancy test at screening or prior to study drug administration.
3. History of significant hypersensitivity to the study drug or excipients of the study drug.
4. History of severe hypersensitivity reactions, such as anaphylaxis.
5. History of rare hereditary problems of galactose and/or lactose intolerance, lactase deficiency or glucose-galactose malabsorption.
6. Positive screening results to HIV antigen and antibody, HBsAg or HCV tests.
7. Poses a significant suicidal risk as defined by C-SSRS score >Type 1 ideation at screening.
8. Any clinically significant illness in the 28 days prior to study drug administration.
9. Presence or history of significant gastrointestinal, liver or kidney disease, or surgery that may affect drug bioavailability.
10. History of significant and uncontrolled or unstable cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic or dermatologic disease.
11. History of seizures (epilepsy) of any kind.
12. History of cranial surgery.
13. Presence of clinically significant ECG abnormalities at the screening visit, as defined by medical judgment (maximum Fridericia's corrected QT interval [QTcF] 450 msec).
14. Any other clinically significant abnormalities in laboratory test results at screening that would, in the opinion of an investigator, increase the subject's risk of participation, jeopardize complete participation in the study, or compromise interpretation of study data. Mild elevations in aspartate aminotransferase (AST)/alanine aminotransferase (ALT) as may be seen in non-alcoholic fatty liver disease (NAFLD) are not exclusionary. However, in these subjects, please follow the hepatic safety section.
15. New prescription medication or changes to medication regimen within 90 days prior to the first dose. (i.e., stable doses of anti-hypertensives etc. are allowed).
16. Use of the following medications for the time frames specified below, with the exception of medications exempted by the Investigator on a case-by-case basis because they are judged unlikely to affect the PK profile of the study drug or subject safety (e.g., topical drug products without significant systemic absorption):

    1. Any vaccination, including COVID-19 vaccine, within 14 days prior to the first dose;
    2. Depot injection or implant of any drug within 3 months prior to the first dose;
    3. Any drugs known to induce or inhibit hepatic drug metabolism within 30 days prior to the first dose.
    4. Any drugs for the treatment of diabetes within 30 days prior to the first dose.
    5. Any drugs prohibited by the Investigator on a case-by-case basis because they are judged likely to affect the PD profile of the study drug or subject safety, within at least 5 times the half-life of the drug and a minimum of 30 days prior to the first dose.
17. Positive urine drug screen or alcohol breath test at screening.
18. History of significant alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to the screening visit (more than 14 units of alcohol per week [1 unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol]).
19. History of significant drug abuse within 1 year prior to screening, use of soft drugs within 3 months prior to screening, marijuana within 1 month prior to screening, or hard drugs (such as cocaine, phencyclidine [PCP], crack, opioid derivatives including heroin, and amphetamine derivatives) within 1 year prior to screening.
20. Use of any cannabinoid containing product, including cannabis, within 1 month prior to screening, by any route (e.g., oral, inhaled, topical).
21. Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days (or a minimum of 5 half-lives, whichever is longer) prior to the first dose, administration of a biological product in the context of a clinical research study within 90 days prior to the first dose, or concomitant participation in an investigational study involving no drug or device administration.
22. Donation of plasma within 7 days prior to dosing. Donation or loss of blood (excluding volume drawn at screening) of 50 mL to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to the first dose.
23. Any reason, which in the opinion of the Investigator, would prevent the subject from participating in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-09-11 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Number and Frequency of Adverse Events | 28 Days
  Safety and Tolerability as assessed by Adverse Events

SECONDARY OUTCOMES:
Pharmacokinetic profile of INV-202 | 28 Days
  Pharmacokinetic profile of INV-202 in blood. Minimum concentration in blood after 1,2,3,and 4 weeks of dosing.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Syneos Health Clinique Inc, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No